CLINICAL TRIAL: NCT05877430
Title: Phase 1/2 Open Label, Safety and Preliminary Efficacy Study of a Live Biotherapeutic Product (CJRB-101) in Combination With Pembrolizumab in Subjects With Selected Types of Advanced or Metastatic Cancer
Brief Title: Safety, Tolerability, and Preliminary Efficacy of CJRB-101 With Pembrolizumab in Subjects With Selected Types of Advanced or Metastatic Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CJ Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CJB-101-01
Record Dates: First submitted 2023-03-12; First posted 2023-05-26 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-08

CONDITIONS: NSCLC; HNSCC; Melanoma; Metastatic Cancer; Advanced Solid Tumor; Advanced Cancer
Keywords: Live Biotherapeutic Product; Keytruda; CJRB-101; metastatic; Immune checkpoint inhibitor; Pembrolizumab; CJB-101-01; anti-PD1; anti-PDL1
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Melanoma; Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CJRB-101 with pembrolizumab (Experimental): Phase 1 includes patients with selected types of advanced or metastatic cancers. Patients will be given with either low or high dose levels of CJRB-101 in combination with pembrolizumab.
  Phase 2 includes patients with selected types of advanced or metastatic cancers. Patients will be given with the CJRB-101 dose selected from Phase 1 in combination with pembrolizumab.
  Interventions: Drug: CJRB-101; Drug: Pembrolizumab injection

INTERVENTIONS:
Drug: CJRB-101 — In Phase 1, one or two capsules of CJRB-101 will be given every day. In Phase 2, the CJRB-101 dose selected from Phase 1 will be given every day.
Drug: Pembrolizumab injection — 200 mg given by intravenous (IV) infusion once every 3 weeks

SUMMARY:
Study CJB-101-01 will be conducted at multiple centers in the USA and Republic of Korea as an open-label safety and preliminary efficacy study of CJRB-101 in combination with pembrolizumab in subjects with selected types of advanced or metastatic cancer. The proposed study intends to address the unmet medical needs of low response rate and refractoriness to immune checkpoint inhibitors typically observed in this subject population by performing assessments of response, dose limiting toxicities, pharmacodynamic, and the effect on microbiome biomarkers at different dose levels of CJRB-101 combined with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent
2. ≥18 years of age at the time of signing the informed consent form
3. Pathologically documented histological or cytological evidence of NSCLC, HNSCC, or melanoma.
4. Has at least 1 measurable target lesion per RECIST v1.1 that has not been resected/biopsied/or irradiated before enrollment in the study
5. Diagnosis of locally advanced unresectable or metastatic NSCLC, HNSCC, or melanoma in subjects who are ICI treatment-naive or relapsed/refractory, including PD-1/PD-L1 inhibitors
6. ICI treatment-naive subjects must meet the following criteria:

   1. NSCLC: Subjects with metastatic or with unresectable, recurrent NSCLC whose tumors must have no EGFR or ALK genomic aberrations and express PD-L1 [TPS≥50%]
   2. HNSCC: Subjects with metastatic or with unresectable, recurrent HNSCC whose tumors express PD-L1 [CPS ≥20]
   3. Melanoma: Irrespective of PD-L1 result and BRAF V600 mutation
   4. Subjects has not received prior systemic treatment for their metastatic tumor. Subjects who received adjuvant or neoadjuvant therapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 6 months before the development of metastatic disease.
7. ICI treatment-refractory subjects as defined by the following criteria:

   1. Has received at least 2 cycles of anti-PD-(L)1 therapy either as monotherapy or in combination
   2. Has demonstrated disease progression after ICI treatment by RECIST v1.1
   3. Has received less than three lines of systemic therapy for metastatic tumor
8. ECOG performance status of 0 or 1
9. Be willing to provide archival tissue or fresh biopsy
10. Have adequate organ function
11. All Grade 3 or greater AEs resolved earlier to Grade 2 or less

Exclusion Criteria:

1. Cancer type and genomic tumor aberrations:

   1. NSCLC subjects with EGFR or ALK genomic tumor aberrations
   2. HNSCC subjects with nasopharyngeal cancer
2. For ICI refractory/relapsed subjects: Immune related AEs ≥Grade 3 that led to discontinuation of prior immune-modulatory agents including PD-1/PD-L1 inhibitors
3. With uncontrolled or untreated brain metastasis or leptomeningeal disease
4. Active autoimmune disease that has required systemic treatment in the past 2 years
5. Received a fecal transplant
6. Concurrent participation in another interventional clinical study or use of another investigational agent within 30 days of study consent
7. Contraindication to IV contrast that cannot be managed with pre-medication
8. Female subjects who are pregnant or breastfeeding
9. Male subjects who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy
10. Has a known inability for oral intake of capsules
11. Has received a live vaccine within 4 weeks of start of the study treatment
12. Diagnosis of prior immunodeficiency or organ transplant requiring immunosuppressive therapy
13. Has received whole blood transfusion, blood component transfusion, or colony stimulating factors within 1 week prior to the 1st dose of study treatment
14. In the judgment of the investigator, subjects unlikely to comply with study procedures, restrictions and requirements
15. Has active interstitial lung disease (ILD)/pneumonitis or a history of ILD/pneumonitis requiring treatment with systemic steroids
16. Have allergy to clindamycin, erythromycin, and ampicillin
17. Has signs and symptoms of colitis at screening
18. Infection requiring systemic antibacterial, antifungal, or antiviral therapy within 14 days before study treatment (Note: Antiviral therapy is permitted for subjects with chronic HBV or HCV infection)
19. Untreated chronic hepatitis B or chronic HBV carriers with HBV DNA>500 IU/mL (or >2500 copies/mL) at screening (Note: Inactive hepatitis B surface antigen (HbsAg) carriers, treated and stable hepatitis B (HBV DNA < 500 IU/mL or < 2500 copies/mL) can be enrolled. Subjects with detectable HbsAg or detectable HBV DNA should be managed per treatment guidelines. Subjects receiving antivirals at screening should have been treated for > 2 weeks before study treatment.)
20. With active hepatitis C (Note: Subjects with a negative HCV antibody test at screening or positive HCV antibody test followed by a negative HCV ribonucleic acid (RNA) test at screening are eligible. The HCV RNA test will be performed only for subjects testing positive for HCV antibody. Subjects receiving antivirals at screening should have been treated for > 2 weeks before study treatment.)
21. Known history of HIV infection
22. History of active inflammatory bowel disease with diarrhea believed to be caused by active inflammatory bowel disease in the past 12 months
23. Major surgery for any reason, except diagnostic biopsy, within 4 weeks of study informed consent and or if the subject has not fully recovered from the surgery within 4 weeks of informed consent
24. History of major gastrointestinal surgery
25. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial
26. Currently active, clinically significant cardiovascular disease
27. Known active intravenous drug or alcohol abuse or use of other drugs of abuse
28. Has any contraindication as mentioned in the recent Keytruda, Highlights of Prescribing Information (pembrolizumab)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
[Phase 1&2] Tolerability and Safety: Incidence of Adverse Events | Maximum 2 years
  Assessed per CTCAE v5.0
[Phase 2] Efficacy | Maximum 2 years
  ORR

SECONDARY OUTCOMES:
[Phase 1&2] Effects of therapy on the microbiome biomarkers - Stool | Maximum 2 years
  Fecal samples will be used to analyze gut microbiome using amplicon sequencing and/or whole-genome shotgun metagenomic sequencing.
[Phase 1&2] Effects of therapy on the pharmacodynamic biomarkers - Blood | Maximum 2 years
  Blood samples will be analyzed for the immune profiling and biomarkers of therapy effect.
[Phase 1&2] Effects of therapy on the pharmacodynamic biomarkers - Tumor | Maximum 2 years
  Tumor tissue samples will be analyzed for immune profiling and evaluated for prediction of therapy effectiveness.
Objective Response Rate (ORR) | Maximum 2 years
  Antitumor effect is assessed through tumor image and tumor lesion per RECIST v1.1.
Disease Control Rate (DCR) | Maximum 2 years
  Antitumor effect is assessed through tumor image and tumor lesion per RECIST v1.1.
Duration Of Response (DOR) | Maximum 2 years
  Antitumor effect is assessed through tumor image and tumor lesion per RECIST v1.1.
Progression Free Survival (PFS) | Maximum 2 years
  Antitumor effect is assessed through tumor image and tumor lesion per RECIST v1.1.
Overall survival (OS) | Maximum 2 years

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - University of California, Irvine, Irvine, California
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Severance Hospital, Seoul